CLINICAL TRIAL: NCT05722184
Title: Diagnostic Evaluation Study of the BactInsight Blood Culture System in West-Africa
Acronym: SIMBLE-FIELD
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Reactivos para Diagnóstico, S.L. (Unknown); University Ghent (Other); Université Libre de Bruxelles (Other); Commissariat A L'energie Atomique (Other Government); Centre Hospitalier Universitaire Yalgado Ouédraogo (Unknown); Centre National Hospitalier et Universitaire de Pneumo-Phtisiologie de Cotonou (Unknown); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Other Study IDs: SIMBLE-FIELD
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Bacterial Infections
Keywords: blood culture; diagnostics
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (3):
- CNHU-HKM: BactInsight system compared to BacT/ALERT® 3D
  Interventions: Diagnostic Test: BactInsight blood culture system
- Hôpital Saint Jean de Dieu, Boko: BactInsight system compared to manual blood culture system (visual inspection)
  Interventions: Diagnostic Test: BactInsight blood culture system
- Centre Hospitalier Universitaire Yalgado Ouédraogo: BactInsight system compared to BacTec FX40
  Interventions: Diagnostic Test: BactInsight blood culture system

INTERVENTIONS:
Diagnostic Test: BactInsight blood culture system — A battery-operated measurement device (turbidimeter), which monitors and detects bacterial growth in blood culture bottles based on the turbidity of the culture medium caused by bacterial growth, in combination with optimized blood culture bottles.

SUMMARY:
Diagnosis of bloodstream infections (BSI) is done by sampling blood in blood culture bottles that are checked for growth in the microbiology laboratory. In LRS, microbiology laboratories are however scarce, and BSI cannot be diagnosed, resulting in overuse of antibiotics which fuels AMR. For diagnosis of BSI, so-called manual blood culture (equipment-free) systems are used in LRS, with daily visual inspection for growth. Compared to automates, manual systems are less sensitive, and growth is slower; in addition, training and experience are needed before laboratory staff is competent to detect growth when inspecting the blood culture bottles.

A simplified blood culture system could enable expanded use of blood cultures in LRS and would thus improve BSI treatment. Ongoing research at the Institute of Tropical Medicine, in collaboration with Ghent University has resulted in a novel, simple, cheap, open-access and robust blood culture system, the Bactinsight blood culture system. This system consists of two modules. Firstly, a portable, battery-operated measurement device (turbidimeter), which monitors and detects bacterial growth in blood culture bottles based on the turbidity of the culture medium caused by bacterial growth. Secondly, optimized blood culture bottles have been developed. A second step in blood cultures is the identification of the causing organism. Researchers at LETI (Grenoble, France) have developed a lensfree microscope, which simplifies and expedites identification of the causative organisms, improving patient's diagnosis and more directed antibiotic treatment. The lensfree microscope is an additional module for the Bactinsight blood culture system.

In SIMBLE, the Bactinsight blood culture system will be evaluated against reference systems in two phases. During the optimization phase in Belgium, the performance of Bactinsight turbidimeter + lensfree microscope will be tested in a reference hospital laboratory. In parallel, an in vitro laboratory evaluation of the Bactinsight blood culture system (turbidimeter + blood culture bottles + lensfree microscope) will be done using spiked blood cultures. In the field-testing phase, the ease-of-use, acceptability, adoptability and performance of Bactinsight blood culture system will be evaluated in three hospitals in Benin and Burkina Faso. The blood culture bottles used for this study will be manufactured in a production facility in Benin, that will be installed at the start of the project.

ELIGIBILITY:
Inclusion Criteria:

* With indications for blood culture sampling and for whom collection of a blood culture sample is part of standard clinical practice
* Willing and able to provide written informed consent (assent for minors)

Exclusion Criteria:

* none

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients older then 15 years old presenting themselves with indications for blood culture sampling and for whom collection of a blood culture sample is part of standard clinical practice.
Sampling Method: Probability Sample
Enrollment: 1724 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Time-to-actionable result | Within 8 days
  The paired Wilcoxon signed rank test will be used to compare the location of the distribution of time-to-actionable result measurements between the two groups for those with a positive blood culture result.
  * BactInsight versus manual system: Time-to-actionable result is compared between both groups with the Wilcoxon signed rank test at the 5% significance level.
  * BactInsight versus automated system: The non-inferiority margin equals 12 hours. Non-inferiority is shown if the upper limit of the two-sided 95% confidence interval for the median of the differences from the Wilcoxon signed rank test is lower than 12h i.e. 12 is excluded from the non-parametric confidence interval.

SECONDARY OUTCOMES:
Time-to-detection | Within 8 days
  The paired Wilcoxon signed rank test will be used to compare the location of the distribution of time-to-detection measurements between the two groups for those with a positive blood culture result.
Yield | 2 years
  The McNemar's test will be used to compare the yield between the BactInsight system and the manual reference system at the 5% significance level in order to detect if there is a statistically significant difference between the paired binary data in terms of proportions.
  o The difference in yield between the BactInsight system and the automated system will be compared to a non-inferiority margin of 15%. Non-inferiority is shown if the lower limit of the two-sided 95% confidence interval is larger than -0.15 i.e. if -0.15 is excluded from the confidence interval. A non-inferiority margin of 15% was chosen as reasonable based on clinical and practical arguments.
Diagnostic performance | 2 years
  Sensitivity and specificity will be calculated for the BactInsight system compared to the composite reference standard, based on the combined result from the components tests i.e. the BactInsight and reference system in use.

OTHER OUTCOMES:
Yield - Antibiotic use | 2 years
  Test whether yield differs in case of antibiotic use (yes/no) within 48 hours prior to blood culture sampling: Pearson Chi-square test (or Fisher exact test in case of small sample size).
Yield - V blood sampled | 2 years
  Test whether yield differs with different volumes of blood sampled (e.g. 5-8 ml; 8-10 ml; 10-15 ml): Pearson Chi-square test (or Fisher exact test in case of small sample size).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Barbé, Principal Investigator — Instituut voor Tropische Geneeskunde
Locations (2):
- Benin (2):
  - Hôpital Saint Jean de Dieu de Boko, Boko
  - Centre National Hospitalier et Universitaire Hubert Koutoukou MAGA, Cotonou

IPD SHARING:
Plan to Share IPD: No